CLINICAL TRIAL: NCT03245359
Title: Pain Management After TKA: Comparison of Short- and Long-term Concurrent Saphenous (Adductor Canal) and Posterior Nerve Blocks Using the ON-Q Pump System
Brief Title: Pain Management After TKA: Comparison of Short- and Long-term Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 880424
Record Dates: First submitted 2017-03-07; First posted 2017-08-10 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia, Local; Pain, Postoperative
Keywords: Total Knee Arthroplasty; Intra-articular Analgesia; Bupivacaine Hydrochloride
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Short-term ON-Q (Active Comparator): Single port, select-a-flow pump and ON-Q 750mL ball filled with bupivacaine 0.125% saphenous (adductor canal) nerve block and single port, fixed flow pump and 400mL ON-Q ball with bupivacaine 0.125% wide field posterior knee block to provide analgesia from surgery until medication has been depleted (typically 2-4 days)
  Interventions: Device: Short-term ON-Q; Drug: Short-term ON-Q
- Long-term ON-Q (Experimental): Single port, select-a-flow pump and two 750mL ON-Q balls filled with bupivacaine 0.125% saphenous (adductor canal) nerve block and single port, fixed flow pump and two 400mL ON-Q ball with bupivacaine 0.125% wide field posterior knee block to provide analgesia from surgery up to 7 days post-operative. The second ball for each location will be provided pre-operatively, along with patient education for connection.
  Interventions: Device: Long-term ON-Q; Drug: Long-term ON-Q

INTERVENTIONS:
Device: Short-term ON-Q — single port, select-a-flow pump connected to saphenous nerve block catheter until medication in initial balls are depleted (usually 2-4 days)
  Arms: Short-term ON-Q
Device: Short-term ON-Q — single port, fixed flow pump connected to posterior knee catheter until medication in initial balls are depleted (usually 2-4 days)
  Arms: Short-term ON-Q
Drug: Short-term ON-Q — Bupivacaine 0.125%
  Arms: Short-term ON-Q
Device: Long-term ON-Q — single port, select-a-flow pump connected to saphenous nerve block catheter until day 7 post-operative
  Arms: Long-term ON-Q
Device: Long-term ON-Q — single port, fixed flow pump connected to posterior knee catheter until day 7 post-operative
  Arms: Long-term ON-Q
Drug: Long-term ON-Q — Bupivacaine 0.125%
  Arms: Long-term ON-Q

SUMMARY:
The purpose of this study is to determine if there is any significant difference between using a short-term ON-Q nerve block (which is applied prior to surgery and maintained in place until the medication in the initial balls have been fully used, usually 2-4 days) in comparison to a long-term ON-Q nerve block (which is applied prior to surgery and maintained in place up to seven days after surgery). This study will analyze patient reported levels of pain, range of motion, and narcotic use, as well as investigate whether blood loss, blood thinners, and hemoglobin/hematocrit blood levels influence patient pain levels.

This study will compare patient-reported pain, range of motion and narcotic use in total knee arthroplasty patients who receive the short-term and long-term combination nerve block (saphenous and posterior of the adductor canal and wide-field posterior knee.

DETAILED DESCRIPTION:
Post-operative pain remains one of the patient's greatest concerns after Total Knee Arthroplasty (TKA). Insufficient pain control can delay mobilization and inhibit rehabilitation efforts. Multimodal analgesia, including peripheral nerve block, is recommended for pain relief, and reaching an effective level of pain management, while minimizing opioid side effects, is vital to a patient's recovery and satisfaction of care delivered. The ON-Q pain relief system continually infuses local analgesia for effective pain relief.

This is a prospective, randomized control trial designed to compare the effects of using the short-term and long-term combination ON-Q nerve blocks in connection with TKA surgery. The ON-Q nerve block and pump system provides slowly infused, continuous delivery of a local anesthetic to the surgical site and nerves. The use of concurrent saphenous and posterior knee nerve blocks with the ON-Q system has been adopted as standard procedure at our institute. The study does not involve an alteration to the typical procedures currently being employed. Ultrasound will ensure the accuracy of catheter placement by a regional anesthesiologist.

All consecutive TKA patients who meet study criteria will be recruited for enrollment in the study prior to surgery. Pre-operatively, patients will be asked to complete health questionnaires, assessments to measure reported pain levels and location, and range of motion. Home medications will be reviewed, and hemoglobin/hematocrit blood levels will be recorded. Patients randomized to the long-term group will receive education on how to connect the ON-Q ball/pump to the catheter using a demonstration set to show understanding of the skill. Patients in the long-term group will also receive a 750mL ON-Q ball/pump filled with bupivacaine 0.125% for the select-a-flow saphenous catheter nerve block and a 400mL ON-Q ball/pump filled with bupivacaine 0.125% for the posterior fixed rate catheter nerve block to enable the nerve blocks to last up to the 7 days of treatment.

Post-operatively, blood loss, inpatient hemoglobin/hematocrit levels, pain medications consumed and side effects, range of motion by Physical Therapy, and pain assessments will be recorded. After discharge, patients will receive daily phone calls up to day 7 post-op to collect reported pain scores, pain medications consumed and side effects, signs/symptoms of catheter site infection, and physical therapy or activity for that day. This information, as well as health questionnaires, will also be collected from both treatment groups at the 2-week and 6-week follow-up office visits.

Data will be analyzed at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Able to provide informed consent
* Undergoing elective total knee arthroplasty
* Able to tolerate both short- and long-term ON-Q therapy

Exclusion Criteria:

* Unable to provide informed consent
* History of dementia or mental instability
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Day of Surgery Pain Scores at 6 Weeks. | This will be collected from day of surgery to 6-weeks postoperative
  This study will assess patient reported pain, as determined by results of the Numeric Pain Rating Scale of 0-10 while knee is at rest and with active bending movement to determine if there is a difference between the short- and long-term groups.
Opioid and Analgesic Use | This will be collected daily from day of surgery through day 7 post-operative.
  Concomitant pain medications consumed while still using the ON-Q nerve block system will be documented, in order to identify reduction/increases in patient's opioid consumption trends.
Number of Participants Who Experience Common Opioid and Analgesic Side Effects | This will be collected daily from day of surgery through day 7 post-operative.
  Concomitant pain medication side effects that are commonly experienced while still using the ON-Q nerve block system will be documented, including nausea, constipation or rash.
Patient Range of Motion (degrees) | This will be completed at all inpatient physical therapy sessions on day 1 and 2 post-operative and follow-up office visits at 2 and 6 weeks post-operative.
  Range of motion measured in degrees will be collected. This will be measured by PI and/or Physical Therapy assessments and used to compare whether there is a difference in the participants range of motion between short- and long-term groups.

SECONDARY OUTCOMES:
Quality of Life - SF-12 | This assessment will be collected at 2- and 6-week follow-up office visits.
  Evaluate the patient quality of life through SF-12 assessment score to assess if there is a trending difference between short- and long-term groups.
Quality of Life - EQ-5D-5L | This assessment will be collected at 2- and 6-week follow-up office visits.
  Evaluate the patient quality of life through EQ-5D-5L assessment score to assess if there is a trending difference between short- and long-term groups.

OTHER OUTCOMES:
Number of Participants with Intraoperative Blood Loss (mL) | Conclusion of Surgery
  Intraoperative blood loss in mL will be collected from patient records
Hemoglobin Laboratory Results (grams/deciliter) | Hemoglobin and hematocrit laboratory results will be collected from the patient's pre-operative testing laboratory results (within 30 days before surgery) and from post-operative inpatient laboratory results (within 48 hours post-operative).
  Hemoglobin levels will be collected from patient records
Hematocrit Laboratory Results (Percentage of Concentration) | Hemoglobin and hematocrit laboratory results will be collected from the patient's pre-operative testing laboratory results (within 30 days before surgery) and from post-operative inpatient laboratory results (within 48 hours post-operative).
  Hematocrit levels will be collected from patient records.

CONTACTS AND LOCATIONS:
Overall Officials: J. Dean Cole, M.D., Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No